CLINICAL TRIAL: NCT04882436
Title: Construction of Special Disease Cohort Database and Biological Sample Holographic Database of Severe Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC2020CR010-001
Record Dates: First submitted 2021-03-28; First posted 2021-05-12 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-05

CONDITIONS: Severe Pneumonia; Special Disease Cohort Database; Holographic Library of Biological Samples
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Biospecimen Retention: Samples With DNA — intravenous blood, sputum, urine, bronchoalveolar lavage fluid and pleural effusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe pneumonia: Patients with severe pneumonia

SUMMARY:
The incidence rate and mortality of lung infection are high worldwide. It is a common and frequently occurring disease which seriously threatens human health. Severe pneumonia accounts for 18-36% of all pneumonia. Severe pneumonia has caused serious economic and medical burden. Therefore, it is urgent to carry out the real-world cohort study of severe pneumonia. Big data and sample library will provide useful clinical guidance and scientific research reserves for clinicians. Through further research, we can improve the treatment success rate and reduce the mortality.

The purpose of this study is to provide reliable biological samples and related data information for the relevant basic and clinical trials in the field of severe pneumonia by carrying out the construction of special disease cohort database and biological sample holographic database, and to establish a long-term sharing platform for the transformation of research results into clinical practice, improve the prognosis of severe pneumonia,and provide the evidence for improving the diagnosis and treatment of severe pneumonia suitable for China's national conditions.

ELIGIBILITY:
Inclusion Criteria:

* Recent cough, expectoration or aggravation of original respiratory diseases, with or without purulent sputum / chest pain / dyspnea / hemoptysis
* Fever
* Signs of pulmonary consolidation and / or moist rales
* Peripheral blood leukocytes >10×10^9/L or less than 4×10^9/L, with or without nucleus shifting to the left.
* New patchy infiltration, consolidation of lobes / segments, ground glass opacity or interstitial changes, with or without pleural effusion on chest imagings
* Positive etiological examination
* Age > 18 years old
* Need mechanical ventilation; septic shock need vasoactive drug treatment. Meet one of them.
* ① respiratory rate ≥ 30 beats / min; ② oxygenation index (PaO2 / FiO2) ≤ 250; ③ multilobar infiltration; ④ disturbance of consciousness / disorientation; ⑤ azotemia (BUN ≥ 20mg / dl); ⑥ cytopenia (WBC < 4.0 × 109 / L); ⑦ thrombocytopenia (platelet < 10.0 × 109 / L); Ⅷ low body temperature (T < 36 ℃); Ⅸ hypotension, requiring strong fluid resuscitation. Meet the above three requirements at the same time.

Exclusion Criteria:

● Cannot understand and / or implement the investigation protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of severe pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
clinical outcome of patients with severe pneumonia | day 3, day 7, day 14, day 30, day 180.
  The pneumonia is cured or improved, or the treatment of pneumonia is invalid, or the patient is dead.

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No